CLINICAL TRIAL: NCT00365651
Title: Multi Intervention Approach to Pediatric Overweight and Obesity: A Randomized Control Group Trial
Brief Title: Nutrition and Soccer for Pediatric Overweight and Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Leach Chiropractic Clinic (Other)
Collaborators: Mississippi University for Women (Other); MUW Southern Women's Institute (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEA2006
Record Dates: First submitted 2006-08-15; First posted 2006-08-17 (Estimated); Last update posted 2007-05-21 (Estimated); Status verified 2007-05

CONDITIONS: Obesity; Overweight
Keywords: obesity; overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Youth Soccer

SUMMARY:
This study will examine whether two months of youth soccer, combined with a single brief behavioral/nutritional intervention, can reduce BMI in 5th grade overweight or obese females.

DETAILED DESCRIPTION:
Female overweight and obese public school students will be recruited during the summer of 2006 based on FitnessGram testing done by graduate students at MSU during their prior (4th grade) school year. After receiving informed consent from parent/child, the subjects will be checked for height/weight and other screening criteria, then exposed to 2005 My Pyramid for Kids, "Tips for Families" information, and watch a short 8 minute DVD that discusses the importance of exercise and fitness by way of interviewing two club level female soccer players of equivalent age. Subjects will then be randomly assigned to fall youth soccer in Starkville, or spring youth soccer, after first phase data collection occurs in November, 2006.

ELIGIBILITY:
Inclusion Criteria:

* obese or overweight 4th grade public school student in Starkville

Exclusion Criteria:

* unable to run or physical disease or disability

Ages: 9 Years to 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2006-06; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
BMI | 5 months

SECONDARY OUTCOMES:
My Tips for Families Quiz | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Leach, DC, MS(c), Principal Investigator — Leach Chiropractic Clinic, Inc; Joyce M Yates, Ed.D., Study Chair — Mississippi University for Women
Locations (1):
- Leach Chiropractic Clinic, Inc., Starkville, Mississippi, United States